CLINICAL TRIAL: NCT01737138
Title: Safety and Effectiveness Study of Percutaneous Catheter-based Renal Sympathetic Denervation in Patients With Chronic Kidney Disease and Resistant Hypertension
Brief Title: Renal Sympathetic Denervation in Patients With Chronic Kidney Disease and Resistant Hypertension
Acronym: RSD4CKD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Qijun Shan, Professor，Director, Cardiac Arrhythmia Group, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-SR-142
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Kidney Disease
Keywords: Resistant hypertension; All-cause mortality; Renal function
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Dosage Forms; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RSD+Medicine (Active Comparator): The investigators will recruit 50 randomised CKD patients who meet the inclusion criteria. First undergo renal artery angiography procedure to confirm anatomy. If renal artery meet the inclusion criteria, give the renal sympathetic denervation. At the same time, we will use optimal medication to protect renal function. Then we will conduct a clinic follow-up and a telephone follow-up e(Total 36 months).
  Interventions: Procedure: RSD
- Medicine (Placebo Comparator): The investigators aslo will recruit 50 randomised CKD patients who meet the inclusion criteria. There are no significant differences in age, gender, race, past medical history,personal history and so on between the two groups. In this group we will use optimal medication just like the RSD+Medicine group. Third we will conduct a clinic and a telephone follow-up(Total 36 months).
  Interventions: Drug: medicine

INTERVENTIONS:
Procedure: RSD — Contrast renal angiography(iodixanol) was performed to localize and assess the renal arteries for accessibility and appropriateness for RSD. Once the anatomy was deemed acceptable, the internally irrigated radiofrequency ablation catheter(Celsius Thermocool,Biosense Webster, Diamond Bar, California) was introduced into each renal artery. then was maneuvered within the renal artery to allow energy delivery in a circumferential, longitudinally staggered manner to minimize the chance of renal artery stenosis. About six to nine ablations at 10 W for 1 min each were performed in both renal arteries. During ablation, the catheter system monitored tip temperature and impedance, altering radiofrequency energy delivery in response to a predetermined algorithm.
  Other Names: renal sympathetic denervation; renal denervation; renal ablation
  Arms: RSD+Medicine
Drug: medicine — Angiotensin converting enzyme inhibitors, angiotensin receptor antagonist, calcium antagonists, diuretic, beta adrenoceptor blocking agent, statins, platelet aggregation inhibitor, anticoagulants and so on.
  Other Names: drug
  Arms: Medicine

SUMMARY:
To study whether renal sympathetic denervation(RSD) is safe and effective in patients with chronic kidney disease and resistant hypertension

DETAILED DESCRIPTION:
Chronic kidney disease(CKD) is a global and growing public health problem, and its frequency increases with age. The major complications of CKD involve losing renal function and cardiovascular disease, which result in significant morbidity, mortality, and cost. The main measures for treatment of CKD are optimizing drug therapy and renal replacement therapy. Optimizing drug therapy, including vascular angiotensin-converting enzyme inhibitors, calcium antagonists, diuretic, beta adrenoceptor blocking agent, statins, platelet aggregation inhibitor, anticoagulants and so on. However, the situation for treatment of CKD is not satisfying. Sympathetic overactivity plays a key role in the development and progression of CKD. Sympathetic nerve activity was increased in patients with all stages of CKD, which was associated with cardiovascular events and all-cause mortality. At the same time, hypertension and proteinuria become the most important risk factor for progression of CKD. Recently, many clinical researches have verified that Catheter-based renal sympathetic denervation can safely be used to substantially reduce muscle and whole-body sympathetic-nerve activity (MSNA) and whole-body norepinephrine spillover. Simultaneously, a marked reduction in blood pressure, sleep apnea severity and urine micro albumin level is apparent, with a improvement glucose tolerance. Sympathetic activation, high norepinephrine level, hypertension, glucose tolerance abnormity, proteinuria and obstructive sleep apnea are all recognized as independent risk factors for the development and progression of CKD. So, we design this randomized parallel control clinical study to demonstrate whether RSD can slow the progression of CKD and reduce the rate of all-cause mortality effectively and securely.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 and ≤75 years of age.
2. A serum creatinine level of 1.5 to 5.0 mg per deciliter (133 to 442 μmol per liter), a creatinine clearance of 20 to 70 ml per minute per 1.73 m2, with variations of less than 30 percent in the three months before randomization.
3. Persistent proteinuria (defined by urinary protein excretion of more than 0.3 g per day for three or more months which can evacuate urinary tract infection and overt heart failure [a New York Heart Association class of III or IV]).
4. Resistant hypertension.
5. Nondiabetic renal disease.
6. Subject is willing and able to comply with the protocol
7. Subject is expected to remain available for follow-up visits at the study center
8. Subject Informed Consent.

Exclusion Criteria:

1. Current treatment with corticosteroids, nonsteroidal antiinflammatory drugs, or immunosuppressive drugs.
2. Connective-tissue disease.
3. Obstructive uropathy.
4. Congestive heart failure (New York Heart Association class III or IV).
5. Subject has significant renovascular abnormalities (a history of prior renal artery intervention, including balloon angioplasty or stenting; double renal artery on one side, distortion, and extension ), measured by abdominal ultrasound or renal angiograms.
6. Subject has a history of myocardial infarction, unstable angina, cerebrovascular accident or alimentary tract hemorrhage in the previous 3 months.
7. Subject with sick sinus syndrome.
8. Subject has a history of allergy to contrast media; psychiatric disorders; drug or alcohol abuse; and pregnancy.
9. Enrolled in a concurrent study that may confound the results of this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-11; Primary Completion 2017-08 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality, doubling of the serum creatinine level or end-stage renal disease | 36 months
  To study the effect of renal sympathetic denervation(RSD) on all-cause mortality,doubling of the serum creatinine level or end-stage renal disease in patients with chronic kidney disease and resistant hypertension.

SECONDARY OUTCOMES:
Urinary protein excretion and renal function | 36 months
  To evaluation of urinary protein excretion and renal function over time, by the reciprocal of the serum and urinary creatinine level, creatinine clearance and the glomerular filtration rate.
Blood pressure | 36 months
  To study the effect of renal sympathetic denervation on blood pressure in patients with hypertension, which can be measured by ambulatory blood pressure and home blood pressure monitoring.
Blood sugar | 36 months
  In order to study whether RSD can reduce the blood sugar level and insulin resistance of diabetic patients. It will be measured by fasting blood glucose, glycated hemoglobin, fasting insulin .
Cardiac function and structure | 36 months
  The effect of renal sympathetic denervation(RSD) on cardiac function and structure can be measured by echocardiographic(include the degree of cardiac pachynesis, left ventricular ejection fraction，left ventricular end diastolic diameter, ventricular septal thickness and so on).
Arrhythmia | 36 months
  If a new arrhythmia is discovered during the follow-up, it will be recorded. Patients may have symptoms of flustered, palpitations, dizziness, amaurosis, syncope and so on, which can be diagnosed by ECG and Holter.
Pulse wave velocity | 36 months
  So as to study whether RSD can improve the patients' blood vessel elasticity, a pulse wave velocity (PWV)will be carried on.
Life quality | 36 months
  Life quality on 36-item short-form(SF-36),HRQoL and PRODISQ Health Survey Questionnaire will be carried out during the follow-up to study the patients' life quality.
Rehospitalization rate | 36 months
  To study whether RSD can reduce the patients' rehospitalization rate, which will be measured by questionnaire and telephone follow-ups.

OTHER OUTCOMES:
Dialysis | 36 months
  In order to study the effect of renal sympathetic denervation on renal function in patients with dialysis, which can be measured by the proportion of patients who do not need dialysis anymore.

CONTACTS AND LOCATIONS:
Overall Officials: Shan Qi Jun, professor, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China